CLINICAL TRIAL: NCT03302884
Title: Circulating Tumor DNA as an Early Marker of Recurrence and Treatment Efficacy in Ovarian Carcinoma
Acronym: CIDOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CIDOC-IPC- 2016-008
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological sampling in ovarian carcinoma (Experimental): Blood and tumor samples
  Interventions: Other: biological sampling

INTERVENTIONS:
Other: biological sampling — Tumor and blood samples

SUMMARY:
Prospective multicentre assay to assess ctDNA value for ovarian cancer monitoring and disease recurrence after front-line treatment.

DETAILED DESCRIPTION:
The main objective is to explore the capacity of ctDNA to be an early marker of ovarian carcinoma recurrence after front-line treatments, i.e. to show significant modifications before clinical diagnosis of disease relapse.

Prospective multicentre open-label study

During visits in the frame of management of the disease, blood samples will be collected at diagnosis, after each cycle of eventual neoadjuvant chemotherapy, every 6 months during the following 2 years, and every year during the remainin time of follow-up. Tumor samples will be collected at surgery or through a biopsy.

Patients will then have a standard care follow-up for a period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with suspicion of ovarian or tubar epithelial cancer, or peritoneal primitive carcino-ma, without previous treatment for ovarian malignancy.
2. Indication of preoperative and/or adjuvant chemotherapy.
3. Age ≥ 18 years old.
4. Patient affiliated to the ''National security'' regimen or beneficiary of this regimen
5. Signed written informed consent prior to any screening procedures being performed

Non inclusion Criteria:

1. Contraindication to surgical assessment.
2. Pathological diagnosis of mucinous carcinoma.
3. History of concurrent malignancy or malignancy within 5 years before study enrollment, (with the exceptions of adequately treated non melanomatous skin cancer or curatively re-sected noninvasive cervical cancer).
4. Assessment by the investigator as being unable or unwilling to comply with the require-ments of the protocol.
5. Patient in urgency situation, adult under legal protection, or unable to give his consent.

Exclusion Criteria after histological exam:

Any diagnostic that is not ovarian or tubar epithelial cancer, or peritoneal primitive carcinoma.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Prognostic value of ctDNA increase for predicting a subsequent clinical, radiological (RECIST v1.1) or biological (CA-125 according to GCIG criteria) diagnosis of disease relapse. | at diagnosis, after each cycle of eventual neo-adjuvant chemotherapy, before surgery, then every six months during the next two years, and every year in the following three years
  Re-appearance of mutations non detectable after treatment or increase of ctDNA comparing to the nadir

CONTACTS AND LOCATIONS:
Overall Officials: Renaud SABATIER, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (3):
- France (3):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - Institut Du Cancer de Montpellier, Montpellier

REFERENCES:
- See also: Description official web site of the sponsor — http://www.institutpaolicalmettes.fr